CLINICAL TRIAL: NCT00369083
Title: Home Hospitalizationfor Elderly Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease: a Randomized Controlled Trial.
Brief Title: Hospitalization at Home of Elderly Patients With Exacerbated COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 515
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2004-01

CONDITIONS: COPD Exacerbation
Keywords: Frail elderly; Hospital at home

INTERVENTIONS:
Procedure: Hospital at home treatment

SUMMARY:
Aim of the study was to evaluate the efficacy of hospital-at-home treatment compared with inpatient care in selected elderly patients with acute exacerbation of chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
A total of 104 patients with an exacerbation of chronic obstructive pulmonary disease (COPD) selected from the Emergency Department (ED) of the hospital were randomized to home treatment from a Geriatric Home Hospitalization Service (GHHS) or to General Medical Ward (GMW).

The sample size estimation was performed according to the increasing 1-year (June 2002-May 2003) incidence of COPD exacerbation in hospital at home. On this basis, al least 100 patients needed to be included in the study to allow to detect a 20% difference in the endpoint hospital iatrogenic diseases, with a statistical significance  = 0.05 and a power 1-  = 0.8 using a two-sided test.

This study is considered a single-blind study because patients were aware of the treatment assignment while physicians and nurses evaluating patients were blinded to the patient's allocation.

In the ED all patients underwent baseline standard clinical evaluation; blood tests (blood cell count, routine biochemical tests and arterial blood gas tensions); pulse oximetry; 12-lead electrocardiography; chest radiographs and hand-held spirometry (SpirHOMEter, COSMED, Italy). Further investigations (including pneumologist's assessment) were performed when required, according to the clinical judgement of the ED physician. Only patients with a COPD exacerbation evaluated in ED for at least 12-24 hours and with stable clinical conditions were considered elegible to be included in the study.

Additional exclusion criteria were: 1) living outside the hospital catchment area; 2) absence of family and social support; 3) absence of informed consent; 4) necessity of intensive monitoring or mechanical ventilation; 5) history of dementia; 6) severe renal or hepatic failure; 7) cancer.

Patients fullfilling inclusion criteria were informed about the nature of the study and asked to give their informed consent. Extensive information was also provided to patients' relatives to obtain their collaboration. Patients fullfilling the inclusion criteria and having none of the criteria for exclusion were randomised, using a set of computer-generated random numbers, in a 1:1 ratio either to the treatment group (home-based hospitalization (GHHS)) or to the control group (conventional care (GMW)), using blinded sealed envelopes. Intention-to-treat analysis was used.

ELIGIBILITY:
Inclusion Criteria:

* Exacerbation of COPD
* Age >= 75 years
* Living in hospital catchment area
* Informed consent
* Adequate social or familial support

Exclusion Criteria:

* Patients requiring assisted ventilation or intensive monitoring
* History of dementia
* Severe renal or hepatic failure
* Cancer

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100
Dates: Start 2004-04; Study Completion 2005-10

PRIMARY OUTCOMES:
Mortality
Hospital readmissions at six months

SECONDARY OUTCOMES:
Length of hospital admission
Caregiver stress
Costs
Patient's quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Aimonino Ricauda, MD, Principal Investigator — San Giovanni Battista Hospital, Torino